CLINICAL TRIAL: NCT00132678
Title: A Randomized, Double-blind, Placebo-controlled Study to Explore the Efficacy and Safety of Risperidone Long-acting Intramuscular Injectable in the Prevention of Mood Episodes in Bipolar 1 Disorder, With Open-label Extension
Brief Title: A Study of the Safety and Efficacy of Injectable Risperidone in the Prevention of Bipolar Mood Episodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR002278; RISBIM3003
Record Dates: First submitted 2005-06-30; First posted 2005-08-22 (Estimated); Results first posted 2009-02-27 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Bipolar Disorder
Keywords: Mood episodes; Bipolar 1 disorder; Intramuscular Injectable; risperidone; safety and efficacy
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Risperdal Consta 12.5 25 37.5 or 50mg intramuscular (IM) injection every 2 weeks
  Interventions: Drug: Risperdal Consta
- 002 (Placebo Comparator): Placebo Matching placebo intramuscular (IM) injection every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperdal Consta — 12.5, 25, 37.5 or 50mg intramuscular (IM) injection every 2 weeks
  Arms: 001
Drug: Placebo — Matching placebo intramuscular (IM) injection every 2 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to determine if risperidone is effective and safe in the prevention of mood episodes in patients with bipolar 1 disorder.

DETAILED DESCRIPTION:
RISPERDAL CONSTA (risperidone long-acting injection) may provide substantial improvement, by reducing patient non-compliance, in the long-term treatment of bipolar I disorder. This is a randomized (patients are assigned different treatments based on chance), double-blind, (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage) placebo-controlled study to explore the safety and effectiveness of RISPERDAL CONSTA in the prevention of mood episodes in patients with bipolar 1 disorder. This study includes 5 periods: a screening period lasting up to 1 week; an open-label RISPERDAL (oral risperidone) treatment period lasting 3 weeks; an open-label RISPERDAL CONSTA stabilization period lasting 26 weeks; a double-blind period lasting up to 24 months; and an open-label extension with RISPERDAL CONSTA lasting 8 weeks. Efficacy will be assessed using the Young Mania Rating Scale (YMRS), Montgomery-Åsberg Depression Rating Scale (MADRS), Clinical Global Impressions - Severity (CGI-S) scale, Medical Outcomes Study Short Form 36 (SF-36), and the Personal and Social Performance (PSP) scale. Safety will be evaluated throughout the study and includes assessment of adverse events, clinical laboratory tests (including hematology, serum chemistry, blood glucose/lipid profile, prolactin, and urinalysis); electrocardiograms (ECGs), vital signs (pulse and blood pressure), physical examination, body mass index (BMI), and the Extrapyramidal Symptom Rating Scale (ESRS). Oral risperidone (flexible dosage) 1 to 6 mg/day for the first 3 weeks. Risperidone LAI i.m. injections (12.5mg, 25 mg, 37.5 mg, or 50 mg) given every 2 weeks for up to approximately 2.6 years (only 6 months for patients receiving placebo during DB-period)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar 1 disorder, currently experiencing a mixed or manic episode or stable
* Two or more bipolar mood episodes in the last 2 years excluding current episode
* Negative pregnancy test

Exclusion Criteria:

* History of > than 4 mood episodes a year during the last two years
* patients experiencing a depressive episode
* History of antisocial or borderline personality illness
* Has unstable or serious general medical illness
* Has received medications disallowed by study criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (51):
- United States (14):
  - Little Rock, Arkansas
  - La Mesa, California
  - National City, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Hialeah, Florida
  - Lake Charles, Louisiana
  - Towson, Maryland
  - Clementon, New Jersey
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - DeSoto, Texas
  - Richmond, Virginia
- Neunkirchen, Austria
- India (3):
  - Bangalore
  - Hyderabad
  - Manipal
- Malaysia (3):
  - Johor Bahru
  - Kota Bharu
  - Kuala Lumpur
- Poland (4):
  - Choroszcz
  - Gdansk
  - Swiecie Poland
  - Tuszyn
- Russia (9):
  - Lipetsk
  - Moscow
  - Moscow Region
  - Moscow Russia
  - Nizny Novgorod
  - Saint Petersburg
  - Samara
  - Saratov
  - St-Petresburg
- Slovakia (3):
  - Bratislava
  - Košice
  - Rimavská Sobota
- Spain (2):
  - Barcelona
  - Madrid
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (8):
  - Dnipro
  - Hlevakha
  - Kharkiv
  - Kiev
  - Lviv
  - Odesa
  - Simferopol
  - Vinnitsa

REFERENCES:
- [Derived] Quiroz JA, Yatham LN, Palumbo JM, Karcher K, Kushner S, Kusumakar V. Risperidone long-acting injectable monotherapy in the maintenance treatment of bipolar I disorder. Biol Psychiatry. 2010 Jul 15;68(2):156-62. doi: 10.1016/j.biopsych.2010.01.015. Epub 2010 Mar 15. PMID 20227682
- See also: A study of the efficacy and safety of injectable risperidone in the prevention of bipolar mood episodes — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=27&filename=CR002278_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 559 (440 + 119) subjects received at least one dose of study drug. A total of 440 subjects (acute episode or stable on other antipsychotic) entered period II, 382 subjects completed and entered period III. An additional 119 subjects (stable on risperidone) entered period III directly. Overall 501 (382 + 119) subjects entered period III.
Pre-assignment Details: Subjects with an acute episode or who were stable on another antipsychotic entered Period II; Period II responders entered Period III. Subjects stable on RIS at screening entered Period III directly. Subjects who maintained response and had a stable dose of RIS LAI for the last 8 weeks of Period III were randomized to RIS LAI or placebo(Period IV).
Groups:
- RISPERDAL CONSTA: risperidone long acting injectable (RIS LAI) 12.5, 25, 37.5 or 50 mg intramuscular (IM) injection every 2 weeks
- Placebo: intramuscular (IM) injection every 2 weeks
- Open-Label Oral Risperidone: (flexible dosage) 1 to 6 mg/day for the first 3 weeks
Period: Period II (Open-Label Oral Risperidone)
Arm/Group | RISPERDAL CONSTA | Placebo | Open-Label Oral Risperidone
Started | 0 | 0 | 440
Completed | 0 | 0 | 382
Not Completed | 0 | 0 | 58
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 13
Not completed — Non responder | 0 | 0 | 6
Not completed — Ineligible to continue trial | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 16
Not completed — Physician Decision | 0 | 0 | 1
Period: Period III (Open-Label Stabilization)
Arm/Group | RISPERDAL CONSTA | Placebo | Open-Label Oral Risperidone
Started | 501 | 0 | 0
Completed | 303 | 0 | 0
Not Completed | 198 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Non responder | 107 | 0 | 0
Not completed — Ineligible to continue trial | 5 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Withdrawal by Subject | 49 | 0 | 0
Not completed — Subject non-compliant | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0
Period: Period IV (Double-Blind Treatment)
Arm/Group | RISPERDAL CONSTA | Placebo | Open-Label Oral Risperidone
Started | 154 | 149 | 0
Completed | 117 | 109 | 0
Not Completed | 37 | 40 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Ineligible to continue the trial | 4 | 4 | 0
Not completed — Lost to Follow-up | 6 | 3 | 0
Not completed — Withdrawal by Subject | 14 | 15 | 0
Not completed — Physician Decision | 10 | 14 | 0
Not completed — Subject Non-compliant | 2 | 1 | 0
Not completed — Pregnancy | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- RISPERDAL CONSTA: risperidone long acting injectable (RIS LAI) 12.5, 25, 37.5 or 50 mg IM injection every 2 weeks
- Placebo: IM injection every 2 weeks
- Total: Total of all reporting groups
Arm/Group | RISPERDAL CONSTA | Placebo | Total
Number analyzed (Participants) | 154 | 149 | 303
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.81) | 39.2 (12.40) | 39.2 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 68 | 147
  Male | 75 | 81 | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Mood Relapse.
Description: Mood Relapse was defined as:
  The subject met DSM-IV criteria for a manic, hypomanic, mixed, or depressive episode; or, the subject needed treatment intervention with any mood stabilizer, antipsychotic medication (other than study drug), benzodiazepine (beyond the dosage allowed), or antidepressant medication; or the subject required hospitalization for any bipolar mood episode; or the subject had a YMRS or MADRS score >12 or a CGI-S score >4; or a dose increase, or supplementation with oral risperidone or another antipsychotic or mood stabilizer, was needed in the opinion of the investigator.
Time Frame: 24 months
Population: Intention to treat. 28 subjects from a Good Clinical Practice noncompliant site and 1 site with alleged research misconduct were excluded from efficacy analyses. The median (interquartile range) for time to relapse (d): Risperdal Consta: NA (173, NA) & Placebo: 219 (82, NA) [NA = not available; Risperdal Consta relapse percent < 50% & Placebo <75%]
Measure: Number; unit: Participants
Arm/Group | RISPERDAL CONSTA | Placebo
Number analyzed (Participants) | 140 | 135
Participants
  Relapsed | 42 [173 to NA] | 76 [82 to NA]
  Not Relapsed | 98 | 59
Statistical Analysis 1: Comparison: RISPERDAL CONSTA vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank; Adjusting for country; Hazard Ratio (HR) = 0.40, 95% CI [0.27 to 0.59] — RISPERDAL CONSTA hazard in numerator, placebo hazard in denominator

2. Secondary Outcome: Change in Young Mania Rating Scale (YMRS) Scores.
Description: Measure of mania; score range 0 to 60 (lower score = less severity)
Time Frame: Baseline and Endpoint (last observation carried forward) of 24 month Double-Blind Period IV
Population: Restricted to subjects with paired baseline and visit endpoint (Period IV) data only. Endpoint is the patient's last nonmissing, postbaseline value in Period IV (last observation carried forward technique)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RISPERDAL CONSTA | Placebo
Number analyzed (Participants) | 135 | 133
units on a scale | 2.9 (7.34) | 9.1 (10.78)
Statistical Analysis 1: Comparison: RISPERDAL CONSTA vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with factors for treatment and country and double-blind baseline value as covariate; Mean Difference (Final Values) = -5.9, 95% CI [-8.08 to -3.79], Standard Error of Mean 1.09 — Change in RISPERDAL CONSTA arm minus change in placebo arm

3. Secondary Outcome: Change in Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: Measure of depression; score range 0 to 60 (lower score = less severity)
Time Frame: Baseline and Endpoint (last observation carried forward) of 24 month Double-Blind Period IV
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RISPERDAL CONSTA | Placebo
Number analyzed (Participants) | 135 | 133
units on a scale | 2.8 (6.66) | 4.9 (8.09)
Statistical Analysis 1: Comparison: RISPERDAL CONSTA vs Placebo; Test type: Superiority or Other; p = 0.020, ANCOVA; ANCOVA model with factors for treatment and country and double-blind baseline value as covariate; Mean Difference (Final Values) = -2.0, 95% CI [-3.75 to -0.32], Standard Error of Mean 0.87 — Change in RISPERDAL CONSTA arm minus change in placebo arm

ADVERSE EVENTS:
Groups:
- RISPERDAL CONSTA: Double-blind Period IV. Risperidone long acting injectable (RIS LAI) 12.5, 25, 37.5 or 50 mg intramuscular (IM) injection every 2 weeks.
- Placebo: Double-blind Period IV. Intramuscular (IM) injection every 2 weeks
- Open-Label Oral Risperidone: Open-label Period II. Flexible dosage. 1 to 6 mg/day for the first 3 weeks
- Open Label RISPERDAL CONSTA: Open-label Period III. Risperidone long acting injectable (RIS LAI) 12.5, 25, 37.5 or 50 mg intramuscular (IM) injection every 2 weeks.
Arm/Group | RISPERDAL CONSTA | Placebo | Open-Label Oral Risperidone | Open Label RISPERDAL CONSTA
Serious Adverse Events (participants affected / at risk) | 13/154 | 25/149 | 8/440 | 38/501
Other Adverse Events (participants affected / at risk) | 28/154 | 24/149 | 81/440 | 155/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RISPERDAL CONSTA (N=154) | Placebo (N=149) | Open-Label Oral Risperidone (N=440) | Open Label RISPERDAL CONSTA (N=501)
Depression (Psychiatric disorders) | 5 | 1 | 0 | 10
Bipolar I disorder (Psychiatric disorders) | 3 | 9 | 2 | 12
Mania (Psychiatric disorders) | 3 | 10 | 1 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 1 | 2
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 3
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Accidental death (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RISPERDAL CONSTA (N=154) | Placebo (N=149) | Open-Label Oral Risperidone (N=440) | Open Label RISPERDAL CONSTA (N=501)
Headache (Nervous system disorders) | 11 | 10 | 33 | 28
Sommolence (Nervous system disorders) | 1 | 1 | 24 | 13
Insomnia (Psychiatric disorders) | 12 | 9 | 23 | 66 — Number affected in Open-Label RISPERDAL CONSTA does not include the event of insomnia in the Serious Adverse Event table.
Anxiety (Psychiatric disorders) | 4 | 6 | 6 | 23 — Number affected in Open-Label RISPERDAL CONSTA does not include the event of anxiety in the Serious Adverse Event table.
Agitation (Psychiatric disorders) | 2 | 7 | 5 | 28
Weight increased (Investigations) | 7 | 1 | 3 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days